CLINICAL TRIAL: NCT03625700
Title: Supplementary Oxygen in Surgical and Medical Wards in the Capital Region of Denmark Evaluated by 30-day Mortality, a Retrospective Cohort Study
Brief Title: Supplementary Oxygen in Surgical and Medical Wards Evaluated by 30-day Mortality
Acronym: SOSAM
Status: Completed | Type: Observational
Sponsor: Hannibal Troensegaard (Other)
Responsible Party: Sponsor-Investigator, Hannibal Troensegaard, Primary investigator, University Hospital Bispebjerg and Frederiksberg
Organization: University Hospital Bispebjerg and Frederiksberg (Other)
Other Study IDs: OxyEWS2018
Record Dates: First submitted 2018-07-10; First posted 2018-08-10 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Oxygen Toxicity; Oxygen Deficiency
MeSH Terms: conditions — Hypoxia | interventions — nitrox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypoxia: Patients without chronic obstructive pulmonary disease: blood oxygen saturation <94 % irrespective of supplemental oxygen
  Patients with chronic obstructive pulmonary disease: blood oxygen saturation <88% irrespective of supplemental oxygen
  Interventions: Drug: Oxygen gas
- Normoxia: Patients without chronic obstructive pulmonary disease: blood oxygen saturation 94-98% in combination with supplemental oxygen OR blood oxygen saturation ≥94% without supplemental oxygen.
  Patients with chronic obstructive pulmonary disease: blood oxygen saturation 88-92% in combination with supplemental oxygen OR blood oxygen saturation ≥88% without supplemental oxygen.
  Interventions: Drug: Oxygen gas
- Hyperoxia: Patients without chronic obstructive pulmonary disease: blood oxygen saturation >98% in combination with supplemental oxygen
  Patients with chronic obstructive pulmonary disease: blood oxygen saturation >92% in combination with supplemental oxygen
  Interventions: Drug: Oxygen gas

INTERVENTIONS:
Drug: Oxygen gas — Supplementary oxygen supplied via nasal catheter or oxygen mask during hospital admission.

SUMMARY:
This study evaluates the use and effects of supplementary oxygen in surgical and medical wards on patients admitted to a hospital in the capital region of Denmark. The population will be divided in to three groups according to their oxygenation status. The main outcome will be 30-day mortality, with secondary outcomes being Length of stay, 30-day admission to ICU, 30-day reoperations, 30-day readmission, and peak values within 30-days of C-reactive protein, S-Creatinine, Troponin.

ELIGIBILITY:
Inclusion Criteria:

* Admission date between 1st of January 2014 to 29th of December 2014 on a hospital in the capital region of Denmark
* Age ≥18
* Unique (first) admission in database for either:
* Hip fracture requiring surgery
* Chronic obstructive pulmonary disease in exacerbation
* Acute mycardial infarction
* Open abdominal surgery

Exclusion Criteria:

* No data on saturation within 48 hours after
* Admission (Medical patients)
* Discharge from the post anaesthesia care unit (Surgical patients)
* No data on primary outcome (30-day mortality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study is made up of four main population groups, each group having their specific vulnerabilities, thus making the main outcome (30-day mortality) more likely to occur than in the background population.
  The four groups are:
  1. Patients undergoing laparotomy (open abdominal surgery)
  2. Patients undergoing orthopedic surgery due to hip fracture
  3. Patients admitted to hospital due to chronic obstructive pulmonary disease in exacerbation
  4. Patients admitted to hospital with acute mycardial infarction
Sampling Method: Probability Sample
Enrollment: 11196 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
30- day mortality | 30 days
  Will be reported as a fraction of positives within the exposure group population

SECONDARY OUTCOMES:
Length of stay | 30 days
  Length of hospital stay in days
Organ markers in blood samples | 30 days
  Highest value of C-reactive protein, Troponin and Creatinine within 30 days.
30- day admission to ICU | 30 days
  Will be reported as a fraction of positives within the exposure group population.
30- day readmission | 30 days
  will be reported as a fraction of positives within the exposure group population.

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg og Frederiksberg Hospital, Copenhagen, NV, Denmark

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03625700/Prot_SAP_000.pdf